CLINICAL TRIAL: NCT06461039
Title: Investigation of the Effect of NNC0487-0111 on Pharmacokinetics of an Oral Combination Contraceptive (Ethinylestradiol and Levonorgestrel) and Gastric Emptying in Females of Non-childbearing Potential
Brief Title: A Research Study Looking at How the Compound NNC0487-0111 Works With Birth Control Pills and Affects Emptying of the Stomach in Women Not Able to Become Pregnant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9487-7612; U1111-1300-3685 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Levonorgestrel; Ethinyl Estradiol; Contraceptive Agents; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNC0487-0111 (Experimental): Participants will receive oral dosing of NNC0487-0111 and gradually will escalate from dose 1 to dose 2. The oral NNC0487-0111 treatment will be followed by s.c. NNC0487-0111 treatment with dose escalating from dose 3 to dose 4.
  Interventions: Drug: NNC0487-0111 A; Drug: NNC0487-0111 C; Drug: Levonorgestrel 150 μg + Ethinylestradiol 30 μg (Oral contraceptive OC); Drug: Acetaminophen - 500 mg/15 ml

INTERVENTIONS:
Drug: NNC0487-0111 A — NNC0487-0111 A will be administered subcutaneously.
Drug: NNC0487-0111 C — NNC0487-0111 C will be taken orally.
Drug: Levonorgestrel 150 μg + Ethinylestradiol 30 μg (Oral contraceptive OC) — Levonorgestrel 150 μg + Ethinylestradiol 30 μg (Oral contraceptive OC) will be taken orally.
Drug: Acetaminophen - 500 mg/15 ml — Acetaminophen - 500 mg/15 ml will be taken orally.

SUMMARY:
This study medicine NNC0487-0111 to improve the treatment options for people living with overweight and obesity or with type 2 diabetes. The purpose of the study is to investigate if NNC0487-0111 affects how effective birth control pills are. Participants will take 1-tablet once daily. The study medicine will taken orally for 18 weeks and then study medicine will be injected with a thin needle in a skin fold in the abdomen for 9 weeks.The study will last for about 35 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential.
* Age 18 - 65 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 25.0 and 39.9 kg/m^2 (both inclusive) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Any disorder, unwillingness or inability which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Any contraindications for the use of the oral contraception used in the study according to the Microgynon Product Information.
* Use of prescription medicinal products or non-prescription drugs including any herbal medicine known to interfere with the metabolic CYP pathways, such as hypericum (St. John's Wort), ginseng, garlic, milk thistle, and echinaceae, within 14 days before screening.

Exceptions are routine vitamins, occasional use of acetaminophen, ibuprofen and acetylsalicylic acid, or topical medication not reaching systemic circulation.

* History of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery) or current presence of gastrointestinal implant.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
The area under the ethinylestradiol plasma concentration time curve at steady state | Day 8 and Day 193
  Measured as hours picograms per milliliter (h*pg/mL).
The area under the levonorgestrel plasma concentration time curve at steady state | Day 8 and Day 193
  Measured as hours picograms per milliliter (h*pg/mL).

SECONDARY OUTCOMES:
Maximum ethinylestradiol plasma concentration at steady state | Day 8 and Day 193
  Measured as picograms per milliliter (pg/mL).
Maximum levonorgestrel plasma concentration at steady state | Day 8 and Day 193
  Measured as picograms per milliliter (pg/mL).
The area under the ethinylestradiol plasma concentration time curve at steady state | Day 8 and Day 135
  Measured as hours picograms per milliliter (h*pg/mL).
The area under the levonorgestrel plasma concentration time curve at steady state | Day 8 and Day 135
  Measured as hours picograms per milliliter (h*pg/mL).
Cmax,EE,SS, maximum ethinylestradiol plasma concentration at steady state | Day 8 and Day 135
  Measured as picograms per milliliter (pg/mL).
Cmax,LN,SS, maximum levonorgestrel plasma concentration at steady state | Day 8 and Day 135
  Measured as picograms per milliliter (pg/mL).
AUC1 area under the acetaminophen concentration-time curve following a standardised meal | Day 1 and Day 186
  Measured as hours micro grams per milliliter (h*μg/mL).
AUC2 area under the acetaminophen concentration-time curve following a standardised meal | Day 1 and Day 186
  Measured as hours micro grams per milliliter (h*μg/mL).
Cmax,para, maximum acetaminophen plasma concentration following a standardised meal | Day 1 and Day 186
  Measured as micrograms per milliliter (μg/mL).
AUC3 area under the acetaminophen concentration-time curve following a standardised meal | Day 1 and Day 128
  Measured as hours micro grams per milliliter (h*μg/mL).
AUC4 area under the acetaminophen concentration-time curve following a standardised meal | Day 1 and Day 128
  Measured as hours micro grams per milliliter (h*μg/mL).
Cmax,para, maximum acetaminophen plasma concentration following a standardised meal | Day 1 and Day 128
  Measured as micrograms per milliliter (μg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical Company, Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com